CLINICAL TRIAL: NCT02407184
Title: Potential Restoration of the Infant Microbiome
Acronym: PRIME
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Bello is no longer a PI at the institution. Data analysis was not completed.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-01446
Record Dates: First submitted 2015-03-05; First posted 2015-04-02 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Human Microbiome
Keywords: Microbiota; Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Scheduled C-section (No Intervention): Babies that are scheduled to be born in a hospital via standard C-section procedure.
- Vaginal Delivery (No Intervention): Babies that are born via vaginal delivery, either at home, at a birthing center or hospital. Drugs may be administered during labor.
- Scheduled C-section with Exposure (Experimental): Babies that are scheduled to be born in a hospital via standard C-section procedure, as well as are swabbed with gauze containing their mother's vaginal microbiota just after delivery. The intervention: Newborn exposure to mother vaginal microbiota.
  Interventions: Other: Newborn exposure to mother vaginal microbiota

INTERVENTIONS:
Other: Newborn exposure to mother vaginal microbiota — Babies are swabbed just after delivery with gauze containing their mother's vaginal microbiota.
  Arms: Scheduled C-section with Exposure

SUMMARY:
Understanding the microbiome's important role in human health, the investigators wish to determine how the development of the infant microbiome is impacted by delivery mode, comparing natural vaginal birth to scheduled C-sections. Investigators will look at the oral, nasal, skin, vaginal and fecal bacteria of 78 mothers and their infants from birth to age 1.

DETAILED DESCRIPTION:
Human microbiota play an important role in the functioning of various organs, as well as the education of the immune system. Mammals have evolved to be born non-sterile, covered with the maternal vaginal bacteria that populate the maternal birth canal, as well as to exclusively breastfeed during early development. Unfortunately, these processes are substantially altered with modern Western practices, which may have health consequences. In particular, C-section is associated with an increased risk of immune diseases and allergies. This study explores the effects of exposing neonates to the vaginal environment at birth, perinatal antibiotics, and lactation on the acquisition of new microbial genes during the first year of infant microbiome development.

This study follows 78 babies from healthy mothers (18-40 years old) with uncomplicated pregnancies. The babies are divided into three groups according to their exposure to the vaginal environment at birth:

Group 1: (n-26) Babies born via vaginal delivery.

Group 2: (n-26) Babies born via scheduled C-section without exposure to mother's vaginal bacteria just after birth.

Group 3: (n-26) Babies born via scheduled C-section with exposure to mother's vaginal microbiota just after birth.

Sampling Time Points:

Subjects may join the study at any point during their pregnancy or soon after delivery. If possible, samples of the mother will be obtained three times prior to delivery in the third trimester: at 30, and 4 or fewer days prior to the mother's due date, as well as on the day of birth prior to delivery. If not possible, samples of mothers and babies can be obtained from birth onwards. Samples will be collected from both mother and baby at day 1, day 2 or 3, weekly through the first month, and monthly through the first year. During monthly sampling, a member of the study team will communicate with mothers regularly to assess for any changes in the infant's diet or health between visits.

Body Sites to be Sampled on Mother and Baby:

At each sampling, a total of 6 samples will be taken from the baby (feces, mouth, nose, forehead skin, right forearm skin, right hand skin) and 9 will be taken from the mother (same as for the babies plus right areola, vagina, and breast milk). Sampling will consist of simple swabbing of the designated body sites, as well as the collection of mother's breast milk.

Each time samples are collected, information about the subject's diet, medication and supplement use, sleep, physical activity and overall health will be asked by survey in order to correlate changes in the life of the subject with changes in his/her microbiota.

C-section with Exposure to the Vaginal Environment Procedure:

Mothers who give birth at NYULMC or Bellevue Hospital and comply with the inclusion and exclusion criteria for exposure to maternal vaginal contents can choose to expose their newborn to samples of their vaginal microbiome just after birth. Such mothers will be tested to confirm that their vaginal pH is acidic (pH ≤ 4), which indicates the dominance of lactic acid bacteria. Testing of vaginal pH will be performed using pH paper. These procedures require of the presence of a study member and will only be performed at NYULMC or Bellevue hospitals.

Samples of vaginal bacteria will be collected prior to C-section. A piece of gauze will be placed in the birth canal just after antibiotic administration, and removed just before the caesarian procedure begins. This period will be no longer than 1 hour long. However, any amount of time the gauze is in the birth canal will be sufficient to proceed with the swabbing procedure. Once removed from the mother, the gauze will be stored in a sterile container until birth. Immediately after delivery, a trained study team member will swab the neonate with the gauze at multiple body sites, starting with the mouth, the face, and then subsequently the remainder of his/her body. After the swabbing, the 6 samples normally taken from all newborns will be collected.

ELIGIBILITY:
Inclusion Criteria for ALL subjects:

* Healthy mothers, 18-40 years old with uncomplicated pregnancies delivering at term (37 weeks or later)
* Mothers of any ethnic or social background that can speak, read, and understand English to the extent that they can consent in English OR mothers who do not speak English yet agree to come to an NYU hospital for all sampling.

Additional inclusion criteria for mothers in the C-section with exposure to the vaginal environment group (CS+E):

* Scheduled C-section
* Vaginal pH ≤ 4 at the time of birth (as measured via pH paper)

Exclusion Criteria for ALL subjects:

* Mothers with pre-eclampsia or other serious chronic conditions
* Mothers with complicated pregnancies
* Mothers under 18 years of age or over 40 years of age
* Babies with complications during delivery
* Babies delivered prior to 37 weeks of gestation

Additional exclusion criteria for mothers in the C-section with exposure to the vaginal environment group (CS+E):

* Mothers reported positive to active primary herpes, genital warts, HIV, Group B Streptococcus, gonorrhea, chlamydia, bacterial vaginosis, yeast infection, or trichomoniasis.
* Mothers with vaginal pH > 4 at the time of birth (as measured via pH paper).
* Known positive Group B Strep test results by rectal vaginal swab within five weeks of the scheduled caesarian.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Bacterial diversity of several body sites on mother and baby throughout one year post-birth as measured by the number and type of different bacteria present | Day of Birth; Days 1 and 3; Weeks 1, 2, 3 and 4; Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11; Year 1
  Investigators will first use Illumina to obtain sequences of the bacterial mitochondrial DNA from collected samples. QIIME, LEfSe, and other bioinformatic tools will then be used to calculate the bacterial diversity (richness, relative abundances) in each sample, as well as compare bacterial communities (beta diversity), sourcetracking to determine origin from maternal sites, random forest to classify communities, and other tools to describe the dynamics of the infant microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gloria Dominguez-Bello, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York, New York, United States